CLINICAL TRIAL: NCT03178955
Title: The Effects of Biologic Therapy With Disease Activity and Circadian Rhythm
Brief Title: Circadian RA Study in Rheumatoid Arthritis Subjects
Status: Withdrawn | Type: Observational
Why Stopped: The Investigator decided not to pursue this study.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1023265
Record Dates: First submitted 2017-06-02; First posted 2017-06-07 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum specimens collected for this study will be immediately sent to the UC Davis clinical laboratory for analysis of RH and CRP. From each study visit, 0.5 ml serum will also be stored to potentially use for analyses of additional markers of inflammation such as interleukin-6 (IL-6). Serum samples will be de-identified; therefore only subject ID numbers will be labeled on the vials of serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Etanercept — Circadian activity rhythm parameters will be evaluated for 7 days prior to Enbrel treatment through 7 days after initiation of Enbrel treatment and again 28-35 days after the second Enbrel treatment.
  Other Names: Enbrel

SUMMARY:
Primary objective: To determine the changes in circadian activity rhythms and disease activity in rheumatoid arthritis (RA) patients from pre-treatment to one month after Enbrel initiation.

Secondary objectives:

* To determine if there is an association between changes in circadian rhythm and changes in disease activity in active RA after initiation of Enbrel
* To determine if the changes in circadian activity rhythms are associated with systemic inflammation in RA patients
* To determine changes in traditional sleep quality variables from pre-treatment to one month after Enbrel initiation in RA patients

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic and debilitating disease. However, the symptoms of RA show variation over the course of the day, with worsening symptoms in the morning. This worsening of symptoms in the morning is correlated with an increase in inflammation in the body.

Biologic therapies, such as Enbrel (etanercept), appear to improve energy, pain and quality of life in patients with RA, and these changes may occur before a doctor is able to detect changes during the patient's physical examination. It is possible that a patient's response to biological agents can be rapidly determined by assessing circadian activity (also called "rest-activity circadian rhythms" or RAR).

Currently, wrist actigraphy bands, which are worn for a period of time, can reliably provide information about RAR. Wrist actigraphy bands are small electronic devices worn on the wrist (similar to a watch) that records the subject's level of activity throughout the day. Studies in osteoarthritis and in rheumatoid arthritis have found subjects with joint pain to have significant differences in RAR, and disrupted RAR has been associated with disease activity.

This study will provide information about 24-hour circadian activity rhythms before and after 3-4 weeks of Enbrel treatment in study subjects with active rheumatoid arthritis. The study will assess patients who are starting on Enbrel that has been prescribed by their doctor.

ELIGIBILITY:
Inclusion Criteria:

* 6/28 tender and 6/28 swollen joints (e.g. active rheumatoid arthritis)
* CRP ≥ 1.5mg/L
* Insufficient response or intolerance to ≥1 disease modifying anti-rheumatic drug (DMARD) which must include methotrexate or hydroxychloroquine, or sulfasalazine or leflunomide and at stable dose for 4 weeks
* If taking Glucocorticoids, stable dose from 0-10mg a day for 2 weeks, and remain stable for the 4 week study
* Appropriate to start on a biologic agent for RA, as determined by patient's physician.

Exclusion Criteria:

* Prior use of a biologic agent for 4 weeks prior to the study
* Evidence of positive tuberculosis (TB) test, purified protein derivative (PPD) or Quantiferon or prophylactic treatment instituted 4 weeks before study, or hepatitis B core antibody
* No medical condition that would prevent completion of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will utilized the UC Davis Cohort Discovery Tool to identify patients within the UC Davis healthcare system who meet the inclusion/exclusion criteria. Investigators will then contact the patients' primary care provider and request permission to contact the patient about the study. Investigators will contact potential subjects to determine their interest and complete screenings by phone. Additionally, investigators plan to advertise the study on flyers posted in the hospital and community, as well as online notices on the Center for Musculoskeletal Health website.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-08-16 (Estimated)

PRIMARY OUTCOMES:
change in pseudo F-statistic | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  indicator of overall robustness of circadian rhythm
change in acrophase | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  time of daily peak circadian activity
change in mesor | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  mean circadian rhythm
change in amplitude | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  indicator of strength of circadian rhythm
change in Disease Activity Score (DAS) | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  RA disease severity

SECONDARY OUTCOMES:
change in sleep efficiency as assessed by wrist actigraphy | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  an index of sleep fragmentation, percentage (%) of time spend sleeping after "lights off"
change in general health visual analogue scale (VAS) | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  subject's general health
change in C-reactive protein (CRP) | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  systemic inflammation
change in rheumatoid factor (RF) | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  measures amount of rheumatoid factor present in the blood
change in sleep duration as assessed by wrist actigraphy | 7 days before, 7 days after and 28-35 days after Enbrel treatment
  how long (minutes) the subject sleeps 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Lane, M.D., Principal Investigator — UC Davis Center for Musculoskeletal Health; Katie Stone, Ph.D., Principal Investigator — California Pacific Medical Center Research Institute
Locations (1):
- UC Davis Center for Musculoskeletal Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No